CLINICAL TRIAL: NCT00610441
Title: A Double Blind, Placebo Controlled, Randomized, Two Period 4-Arm Trial to Investigate the Dose-Related Efficacy and Safety of Org 26576 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Dose Finding Study in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)(174007/P05805/MK-8777-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P05805; 174007 (Other: Organon Protocol Number)
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: randomized; double blind; placebo controlled
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-8777 FD→PBO (Experimental): Participants receive a fixed dose (FD) of MK-8777 100 mg twice each day (BID) for 3 weeks (Treatment Period 1). After a 2-week placebo washout period, participants receive a fixed dose of placebo (PBO) BID for 3 weeks (Treatment Period 2).
  Interventions: Drug: MK-8777; Drug: Placebo
- PBO→MK-8777 FD (Experimental): Participants receive a fixed dose of placebo BID for 3 weeks (Treatment Period 1). After a 2-week placebo washout period, participants receive a fixed dose of MK-8777 100 mg BID for 3 weeks (Treatment Period 2).
  Interventions: Drug: MK-8777; Drug: Placebo
- MK-8777 RD→PBO (Experimental): Participants receive rising doses (RD) of MK-8777 100-300 mg BID for 3 weeks (Treatment Period 1). After a 2-week placebo washout period, participants receive rising doses of placebo BID for 3 weeks (Treatment Period 2).
  Interventions: Drug: MK-8777; Drug: Placebo
- PBO→MK-8777 RD (Placebo Comparator): Participants receive rising doses of placebo BID for 3 weeks (Treatment Period 1). After a 2-week placebo washout period, participants receive rising doses of MK-8777 100-300 mg BID for 3 weeks (Treatment Period 2).
  Interventions: Drug: MK-8777; Drug: Placebo

INTERVENTIONS:
Drug: MK-8777
Drug: Placebo

SUMMARY:
This is a Phase 2 multicenter, randomized, double-blind trial of MK-8777 (Org 26576, SCH 900777) in adult subjects with Attention-Deficit/Hyperactivity Disorder (ADHD). MK-8777 or placebo will be administered in a crossover fashion for two 3-week treatment periods. The two 3-week treatment periods will be separated by a 2-week placebo washout period.

The primary objective is to compare the efficacy of various doses of MK-8777 to that of placebo in the treatment of ADHD symptoms in adults.

ELIGIBILITY:
Inclusion Criteria:

* are between 18-50 years, inclusive;
* are male; or female who are non-pregnant, non-lactating and using an acceptable method of birth control (intrauterine device, double-barrier method, hormonal contraceptives); or female of non-childbearing potential if they are a) surgically sterile (tubal ligation, hysterectomy and/or bilateral oophorectomy) and provide documentation of the procedure by operative report or ultrasound scan, or b) post-menopausal for greater than one year with follicle stimulating hormone (FSH) level greater than or equal to 40 mIU/mL at screening. All females must have a negative serum pregnancy test at screening;
* are outpatients;
* provide written informed consent
* are fluent in the language of the investigator,
* are able to discontinue the use of any psychotropic medications for the treatment of ADHD symptoms at screening;
* meet strict operational criteria for adult ADHD according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV-TRTM)
* have a Clinical Global Impression ADHD score of 4 or higher at screening

Exclusion Criteria:

* have any clinically significant concurrent medical condition (endocrine, renal, respiratory, cardiovascular, hematological, immunological, cerebrovascular, neurological, anorexia, obesity or malignancy) that has become unstable and may interfere with the interpretation of safety and efficacy evaluations.
* have any clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram (ECG) findings at screening that, in the opinion of the investigator, may interfere with the interpretation of safety or efficacy evaluations.
* have any history of liver disease (e.g., cirrhosis, hepatitis), or liver injury;(history of hepatitis A greater than one year prior to screening is acceptable); any abnormal clinically significant findings at screening on liver laboratory parameters (serum glutamic-pyruvic transaminase [SGPT], serum glutamic oxaloacetic transaminase [SGOT], gamma-glutamyltransferase [GGT], lactate dehydrogenase [LDH], bilirubin, albumin, protein, alkaline phosphatase);
* have a seizure disorder beyond childhood or are taking any anticonvulsants to prevent seizures;
* have known serological evidence of human immunodeficiency virus (HIV) antibody;
* have a positive test result at screening on hepatitis B surface antigen or hepatitis A immunoglobulin M (IgM) antibodies or hepatitis C total antibodies;
* are pregnant as confirmed by a positive serum pregnancy test at screening;
* have QTc values >450 msec at screening using Fridericia's QTc formula;
* have a confirmed positive result in the alcohol/drug screen test for alcohol, illegal or non-prescribed drugs at screening (except marijuana/ tetrahydrocannabinol [THC]);
* have a confirmed positive result in the alcohol/drug screen re-test for marijuana/THC;
* have current or lifetime history of bipolar and psychotic disorders;
* have a current major depression disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, panic disorder and eating disorder (also if treated but not currently symptomatic);
* have a current comorbid dysthymia or social anxiety disorder that is currently treated with psychotropic medication;
* have a current untreated social anxiety disorder that may interfere with the assessment of ADHD in the investigator's opinion;
* present an imminent risk of self-harm or harm to others;
* have any history of a significant suicide attempt, or possess a current risk of attempting suicide, in the investigator's opinion, based on clinical interview and responses provided on the Beck Scale for Suicidal Ideation (BSS);
* have a history of jailing or imprisonment in the past 6 months due to worsening of symptoms of ADHD;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2009-03-02 (Actual); Study Completion 2009-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-8777 FD→PBO: Participants receive a fixed dose (FD) of MK-8777 100 mg BID for 3 weeks (Treatment Period 1). After a 2-week placebo washout period, participants receive a fixed dose of placebo BID for 3 weeks (Treatment Period 2).
Period: Treatment Period 1 - 3 Weeks
Arm/Group | MK-8777 FD→PBO | PBO→MK-8777 FD | MK-8777 RD→PBO | PBO→MK-8777 RD
Started | 15 | 16 | 18 | 18
Completed | 12 | 14 | 11 | 16
Not Completed | 3 | 2 | 7 | 2
Not completed — Adverse Event | 1 | 1 | 4 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Period: Placebo Washout Period - 2 Weeks
Arm/Group | MK-8777 FD→PBO | PBO→MK-8777 FD | MK-8777 RD→PBO | PBO→MK-8777 RD
Started | 12 | 14 | 11 | 16
Completed | 12 | 13 | 9 | 16
Not Completed | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Treatment Period 2 - 3 Weeks
Arm/Group | MK-8777 FD→PBO | PBO→MK-8777 FD | MK-8777 RD→PBO | PBO→MK-8777 RD
Started | 12 | 13 | 9 | 16
Completed | 10 | 12 | 9 | 14
Not Completed | 2 | 1 | 0 | 2
Not completed — Other | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-8777 FD→PBO: Participants receive a fixed dose FD of MK-8777 100 mg BID for 3 weeks (Treatment Period 1). After a 2-week placebo washout period, participants receive a fixed dose of placebo BID for 3 weeks (Treatment Period 2).
- MK-8777 RD→PBO: Participants receive rising doses of MK-8777 100-300 mg BID for 3 weeks (Treatment Period 1). After a 2-week placebo washout period, participants receive rising doses of placebo BID for 3 weeks (Treatment Period 2).
- Total: Total of all reporting groups
Arm/Group | MK-8777 FD→PBO | PBO→MK-8777 FD | MK-8777 RD→PBO | PBO→MK-8777 RD | Total
Number analyzed (Participants) | 15 | 16 | 18 | 18 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (8.7) | 35.1 (9.2) | 36.7 (8.8) | 40.7 (6.3) | 37.0 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 9 | 5 | 22
  Male | 12 | 11 | 9 | 13 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Investigator Symptom Rating Scale (AISRS) Score
Description: The AISRS is an 18-item clinician-rated instrument for assessing the 18 core symptoms of ADHD corresponding to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnostic symptoms for adults. Based on the clinician's rating for each of the symptoms using a 4-point scale (0=None to 3=Severe), the AISRS total score is derived by summing the score assigned to each of the 18 symptoms. Scores can range from 0 to 54, with a higher score indicating a more severe ADHD symptoms. Baseline was defined as the score at the baseline visit prior to starting dosing for Period 1 and as the last score in the 2-week placebo wash-out period for Period 2. For the statistical analyses, the average score from Day 14 and Day 21 was used.
Time Frame: Baseline (BL) and Day 7, Day 14, Day 21
Population: The Intent-to-Treat (ITT) population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline AISRS efficacy assessment. Results are reported by the study drug being administered at time of assessment and not by randomly assigned sequence.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD; Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD: Participants who received placebo in either Treatment Period 1 or Treatment Period 2.
- MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD: Participants who received a fixed dose of MK-8777 100 mg BID in either Treatment Period 1 or Treatment Period 2.
- MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD: Participants who received rising doses of MK-8777 100-300 mg BID in either Treatment Period 1 or Treatment Period 2.
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 25 | 27 | 27 | 30
score on a scale
  Change from BL at Day 7 (n=25, 26, 27, 30) | 0.0 (6.7) | -3.7 (7.1) | -3.4 (6.5) | -3.9 (7.6)
  Change from BL at Day 14 (n=25, 27, 27, 27) | -1.4 (9.4) | -7.3 (8.6) | -5.1 (7.4) | -4.6 (7.7)
  Change from BL at Day 21 (n=22, 25, 24, 23) | -1.0 (8.9) | -7.5 (10.8) | -6.8 (9.1) | -3.3 (9.4)
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; The treatment difference between 100 mg MK-8777 fixed dose and Placebo was estimated for the average effect (average change from baseline) of the 2nd and 3rd week of each period (Day 14 and Day 21); Test type: Superiority or Other; p = 0.0147, Mixed Model for Repeated Measurements — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = -5.6996, 97.5% CI 2-sided [-10.911 to -0.4881] — Mixed Model for Repeated Measurements (MMRM) with fixed effects for treatment, period, visit, center and treatment by visit interaction, and random effect for participant, and baseline AISRS score as covariate
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; The treatment difference between 100-300 mg MK-8777 rising dose and Placebo was estimated for the average effect (average change from baseline) of the 2nd and 3rd week of each period (Day 14 and Day 21); Test type: Superiority or Other; p = 0.5910, MMRM — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = 0.9926, 97.5% CI 2-sided [-3.2961 to 5.2814] — MMRM with fixed effects for treatment, period, visit, center and treatment by visit interaction, and random effect for participant, and baseline AISRS score as covariate

2. Secondary Outcome: Percentage of Participants With at Least a 30% Reduction From Baseline in AISRS Score
Description: The AISRS is an 18-item clinician-rated instrument for assessing the 18 core symptoms of ADHD corresponding to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnostic symptoms for adults. Based on the clinician's rating for each of the symptoms using a 4-point scale (0=None to 3=Severe), the AISRS total score is derived by summing the score assigned to each of the 18 symptoms. Scores can range from 0 to 54, with a higher score indicating a more severe ADHD symptoms. Baseline was defined as the score at the baseline visit prior to starting dosing for Period 1 and as the last score in the 2-week placebo wash-out period for Period 2. Reduction was defined as the relative change from the baseline score within a treatment period to post-baseline score within that treatment period.
Time Frame: Baseline and Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug, and who had at least one postbaseline AISRS efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 25 | 27 | 27 | 27
percentage of participants | 12.0 | 41.0 | 33.0 | 30.0
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; Test type: Superiority or Other; Odds Ratio (OR) = 6.8506, 95% CI 2-sided [1.7990 to 26.0878] — Logistic regression with fixed effects for treatment and period, and baseline AISRS score as covariate
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; Test type: Superiority or Other; Odds Ratio (OR) = 0.9461, 95% CI 2-sided [0.3119 to 2.8701] — Logistic regression with fixed effects for treatment and period, and baseline AISRS score as covariate

3. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in AISRS Score
Description: The AISRS is an 18-item clinician-rated instrument for assessing the 18 core symptoms of ADHD corresponding to the DSM-IV diagnostic symptoms for adults. Based on the clinician's rating for each of the symptoms using a 4-point scale (0=None to 3=Severe), the AISRS total score is derived by summing the score assigned to each of the 18 symptoms. Scores can range from 0 to 54, with a higher score indicating a more severe ADHD symptoms. Baseline was defined as the score at the baseline visit prior to starting dosing for Period 1 and as the last score in the 2-week placebo wash-out period for Period 2. Reduction was defined as the relative change from the baseline score within a treatment period to post-baseline score within that treatment period.
Time Frame: Baseline and Day 21
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 27 | 27
percentage of participants | 0.0 | 19.0 | 19.0 | 4.0
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; Test type: Superiority or Other; Odds Ratio (OR) = 6.2468, 95% CI 2-sided [0.6712 to 58.1395] — Since no participants in the Placebo group achieved a 50% reduction, the comparison was done using a Cochran-Mantel-Haenszel method and 0.5 was added to both groups
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; Test type: Superiority or Other; Odds Ratio (OR) = 0.1453, 95% CI 2-sided [0.0152 to 1.3880] — Logistic regression with fixed effects for treatment and period, and baseline AISRS score as covariate

4. Secondary Outcome: Percentage of Participants Who Experience At Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not related to the investigational product. AEs are reported by study drug taken at time of event and not by randomly assigned sequence.
Time Frame: Up to 7 days after last dose of study drug (Up to 63 days)
Population: The All-Subjects-Treated (AST) population consisted of all participants who received at least one dose of randomized study drug within at least one of the two treatment periods (excluding the placebo run-in period).
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants receive placebo BID for 3 weeks.
- MK-8777 100mg: Participants receive a fixed dose of MK-8777 100 mg BID for 3 weeks.
- MK-8777 100-300mg: Participants receive rising doses of MK-8777 100-300 mg BID for 3 weeks.
Arm/Group | Placebo | MK-8777 100mg | MK-8777 100-300mg
Number analyzed (Participants) | 55 | 28 | 34
percentage of participants | 56.4 | 71.4 | 85.3

5. Secondary Outcome: Percentage of Participants Who Discontinue Study Drug Due to an AE
Description: as for outcome 4
Time Frame: Up to last dose of study drug (Up to 56 days)
Population: The AST population consisted of all participants who received at least one dose of randomized study drug within at least one of the two treatment periods (excluding the placebo run-in period).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MK-8777 100mg | MK-8777 100-300mg
Number analyzed (Participants) | 55 | 28 | 34
percentage of participants | 3.6 | 3.6 | 20.6

6. Secondary Outcome: Percentage of Participants With Clinician Global Impression Scale - Severity (CGI-S) Category Scores
Description: The CGI-S is a 7-point clinician-rated scale for assessing the global severity of ADHD. Scores could range from 1=Normal, not at all ill to 7=Among the most extremely ill, with a higher score indicating more severe illness. Categorization was as follows: 1=Normal, not at all ill and Borderline mentally ill; 2=Mildly ill; 3=Moderately ill and 4=Markedly ill, Severely ill and Among the most extremely ill patients, with a higher category indicating more severe illness. Analysis of CGI-S was performed using a proportional odds model. For statistical analyses, CGI-S assessments were condensed to one assessment of severity per treatment period by taking the most severe score at the second and third visits within a treatment period.
Time Frame: Days 14-21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug, and who had at least one postbaseline CGI-S efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 28 | 27 | 32
percentage of participants
  Category 1 | 4.00 | 3.70 | 3.70 | 7.41
  Category 2 | 20.00 | 14.81 | 11.11 | 22.22
  Category 3 | 36.00 | 55.56 | 55.56 | 51.85
  Category 4 | 40.00 | 25.93 | 29.63 | 18.52
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; Test type: Superiority or Other; Odds Ratio (OR) = 1.2074, 95% CI 2-sided [0.5654 to 2.5785] — Proportional odds model with fixed effects for treatment and period
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; Test type: Superiority or Other; Odds Ratio (OR) = 1.8548, 95% CI 2-sided [0.6951 to 4.9494] — Proportional odds model with fixed effects for treatment and period

7. Secondary Outcome: Percentage of Participants With Clinician Global Impression Scale - Improvement (CGI-I) Scores
Description: The CGI-I is a 7-point clinician-rated scale for assessing the global improvement of ADHD. Scores could range from 1=Very much improved to 4=No change to 7=Very much worse, with a lower score indicating the most improvement. Analysis of CGI-I was performed using a proportional odds model. For statistical analyses, CGI-I assessments were condensed to one assessment of improvement per treatment period by taking the worst improvement score at the second and third visits within a treatment period.
Time Frame: Days 14-21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug, and who had at least one postbaseline CGI-I efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 28 | 27 | 32
percentage of participants
  Score of 1 | 0.0 | 3.70 | 3.70 | 3.70
  Score of 2 | 12.00 | 11.11 | 3.70 | 14.81
  Score of 3 | 20.00 | 25.93 | 40.74 | 40.74
  Score of 4 | 64.00 | 55.56 | 48.15 | 33.33
  Score of 5 | 4.00 | 3.70 | 3.70 | 7.41
  Score of 6 | 0.00 | 0.00 | 0.00 | 0.00
  Score of 7 | 0.00 | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; Test type: Superiority or Other; Odds Ratio (OR) = 1.3149, 95% CI 2-sided [0.5402 to 3.2008] — Proportional odds model with fixed effects for treatment and period
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; Test type: Superiority or Other; Odds Ratio (OR) = 1.3982, 95% CI 2-sided [0.5240 to 3.7309] — Proportional odds model with fixed effects for treatment and period

8. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Score
Description: The ESS is an 8-item scale used to assess sleepiness. The test consists of a list of 8 situations in which participants rate their tendency to become sleepy on a scale of 0=Would never doze to 3=High chance of dozing. The scores for each of the 8 situations are added to create a total score on a scale with a range from of 0 to 24. A higher score indicates a greater degree of sleepiness. Baseline was defined as the score at the baseline visit prior to starting dosing for Period 1 and as the last score in the 2-week placebo wash-out period for Period 2.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline ESS efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 25 | 27 | 27 | 30
score on a scale
  Change from BL at Day 7 (n=25, 25, 27, 30) | -0.6 (4.0) | -1.1 (2.5) | -0.7 (3.1) | 1.5 (5.4)
  Change from BL at Day 14 (n=25, 27, 27, 27) | -1.6 (3.8) | -1.7 (2.3) | -1.3 (3.7) | 1.2 (4.7)
  Change from BL at Day 21 (n=22, 25, 24, 23) | -0.9 (4.0) | -0.8 (3.8) | -0.7 (4.6) | 1.1 (3.1)
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6155, MMRM — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = -0.3163, 97.5% CI 2-sided [-1.8138 to 1.1812] — MMRM with fixed effects for treatment, period, visit, center and treatment by visit interaction, and random effect for participant, and baseline ESS score as covariate. For statistical analyses, the average score from Days 14 and 21 was used
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1330, MMRM — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = 1.2934, 97.5% CI 2-sided [-0.7449 to 3.3317] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Score
Description: The PSQI is a participant-rated scale to assess the quality of sleep. The PSQI consists of 7 component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component score can range from 0=better (i.e., 0 times per month) to 3=worse (i.e., 3 or more times per week). The sum of these 7 component scores yields one total score with a range of 0 (better) to 21 (worse). A total PSQI score <=5 is associated with good sleep quality; a total score >5 is associated with poor sleep quality. Baseline was defined as the score at the baseline visit prior to starting dosing for Period 1 and as the last score in the 2-week placebo wash-out period for Period 2.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline PSQI efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 25 | 27 | 27 | 30
score on a scale
  Change from BL at Day 7 (N=25, 26, 27, 30) | -0.7 (1.7) | -0.6 (2.0) | 0.6 (3.2) | -0.4 (2.2)
  Change from BL at Day 14 (N=25, 27, 27, 27) | -0.5 (1.7) | -0.1 (3.6) | -0.8 (2.3) | -0.1 (2.4)
  Change from BL at Day 21 (n=21, 25, 24, 23) | -1.1 (2.5) | -0.7 (2.7) | -0.4 (2.1) | -0.3 (2.6)
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3907, MMRM — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = 0.5501, 97.5% CI 2-sided [-0.9427 to 2.0429] — MMRM with fixed effects for treatment, period, visit, center and treatment by visit interaction, and random effect for participant, and baseline PSQI score as covariate
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9872, MMRM — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = -0.0065, 97.5% CI 2-sided [-0.9486 to 0.9357] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Change From Baseline in Quick Inventory of Depression Symptomology - Clinician Rating (QIDS-C) Score
Description: The QIDS-C is a clinician-administered rating scale to measure the severity of depressive symptoms within the 9 DSM-IV major depression disorder symptom (MDD) domains: depressed mood, loss of interest or pleasure, concentration/decision making, self-outlook, suicidal ideation, energy/fatigability, sleep, weight/appetite change, and psychomotor changes. There is one score (0=none to 3=severe) for each of the of the 9 domains. The total score is obtained by adding the scores for each of the 9 symptom domains. QIDS-C total scores can range from 0 to 27, with a higher score indicating more severe depression. Baseline was defined as the score at the baseline visit prior to starting dosing for Period 1 and as the last score in the 2-week placebo wash-out period for Period 2.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline QIDS-C efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 25 | 27 | 27 | 30
score on a scale
  Change from BL at Day 7 (n=25, 26, 27, 30) | 0.2 (1.7) | -0.1 (2.3) | -0.1 (2.2) | -0.3 (2.5)
  Change from BL at Day 14 (n=25, 27, 27, 27) | 0.3 (2.9) | 0.0 (2.9) | -0.3 (1.4) | 0.3 (2.5)
  Change from BL at Day 21 (n=22, 25, 24, 23) | 0.1 (2.6) | 0.5 (2.1) | -0.5 (1.9) | 0.1 (2.7)
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7828, MMRM — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = -0.1543, 97.5% CI 2-sided [-1.4898 to 1.1811] — MMRM with fixed effects for treatment, period, visit, center and treatment by visit interaction, and random effect for participant, and baseline QIDS-C score as covariate. Scores from Days 14 and 21 were averaged for statistical analyses
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2883, MMRM — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = 0.4222, 97.5% CI 2-sided [-0.5187 to 1.3630] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Change From Baseline in Time-Sensitive ADHD Symptom Scale (TASS) Score
Description: The TASS is a participant-administered scale to assess study drug effects in the evening. Participants respond to 18 questions about ADHD symptoms, with scores from 0=Not at all to 3=Severe. Total scores can range from 0 to 54, with a higher score indicating more severe ADHD symtoms. Baseline was defined as the score at the baseline visit prior to starting dosing for Period 1 and as the last score in the 2-week placebo wash-out period for Period 2.
Time Frame: Baseline and Day 7, Day 14, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline TASS efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 20 | 23 | 22 | 25
score on a scale
  Change from BL at Day 7 (n=20, 23, 22, 25) | 0.3 (6.5) | -1.1 (6.5) | 0.0 (6.2) | -1.5 (4.7)
  Change from BL at Day 14 (n=20, 22, 20, 25) | -0.4 (8.1) | -2.2 (7.8) | -2.4 (6.2) | -1.7 (6.5)
  Change from BL at Day 21 (n=15, 23, 21, 19) | -2.2 (7.3) | -3.0 (8.7) | -2.9 (8.4) | -1.3 (6.9)
Statistical Analysis 1: Comparison: Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD vs MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6532, MMRM; To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = -0.9685, 97.5% CI 2-sided [-5.9599 to 4.0229] — MMRM with fixed effects for treatment, period, visit, center and treatment by visit interaction, and random effect for participant, and baseline TASS score as covariate
Statistical Analysis 2: Comparison: Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD vs MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5247, MMRM — To correct for multiplicity, p-values (2-sided) should be compared with the 2.5% level of significance; Mean Difference (Net) = 1.1022, 97.5% CI 2-sided [-2.8951 to 5.0996] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Computerized Cognition Assessment: Cognitive Flexibility
Description: Cognition was assessed by a computerized cognitive testing (©CNS Vital Signs, Chapel Hill, NC) battery consisting of neuropsychological tests that measure the cognitive domain of cognitive flexibility (score range: -200 to 200), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for cognitive flexibility.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 48.0 (18.1) | 49.5 (17.9) | 47.1 (19.5) | 46.5 (20.5)
  Day 21 (n=21, 25, 25, 23) | 50.3 (14.1) | 49.2 (20.7) | 50.9 (14.8) | 50.7 (16.5)

13. Secondary Outcome: Computerized Cognition Assessment: Complex Attention
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of complex attention (score range: 0 to 250), with a lower score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for complex attention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 11.9 (22.0) | 17.3 (32.0) | 13.5 (26.1) | 10.8 (15.9)
  Day 21 (n=21, 25, 25, 23) | 18.1 (39.0) | 12.8 (14.4) | 9.6 (15.5) | 16.0 (31.3)

14. Secondary Outcome: Computerized Cognition Assessment: Composite Memory
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of composite memory (score range: -120 to 120), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for composite memory.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 92.5 (8.7) | 92.6 (10.5) | 96.9 (9.7) | 96.7 (9.4)
  Day 21 (n=21, 25, 25, 23) | 98.8 (10.2) | 93.1 (9.5) | 96.0 (11.8) | 96.0 (12.4)

15. Secondary Outcome: Computerized Cognition Assessment: Executive Functioning
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of executive functioning (score range: -200 to 200), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for executive functioning.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 49.8 (17.1) | 50.9 (17.7) | 49.3 (19.5) | 48.1 (20.3)
  Day 21 (n=21, 25, 25, 23) | 52.0 (13.7) | 50.9 (19.7) | 53.1 (14.0) | 52.5 (15.6)

16. Secondary Outcome: Computerized Cognition Assessment: Speed of Processing
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of speed of processing (score range: -1000 to 200), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for speed of processing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 63.8 (16.1) | 64.3 (15.8) | 58.0 (10.6) | 58.9 (8.0)
  Day 21 (n=21, 25, 25, 23) | 64.1 (9.1) | 63.5 (15.5) | 60.9 (10.6) | 59.9 (9.0)

17. Secondary Outcome: Computerized Cognition Assessment: Reaction Time
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of reaction time (lowest time possible is 0 msec), with a lower reaction time indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for reaction time.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
msec
  BL (n=27, 27, 26, 32) | 646.7 (87.3) | 645.6 (81.6) | 653.1 (118.8) | 673.8 (124.1)
  Day 21 (n=21, 25, 25, 23) | 634.4 (74.6) | 621.7 (152.0) | 646.7 (139.3) | 642.4 (111.5)

18. Secondary Outcome: Computerized Cognition Assessment: Reasoning
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of reasoning (score range: -15 to 15), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for reasoning.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 6.6 (4.6) | 7.7 (4.6) | 5.9 (3.3) | 7.5 (3.3)
  Day 21 (n=21, 25, 25, 23) | 7.9 (3.3) | 8.2 (3.7) | 7.4 (4.1) | 7.1 (3.7)

19. Secondary Outcome: Computerized Cognition Assessment: Sustained Attention
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of sustained attention (score range -120 to 120), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for sustained attention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 26.1 (12.0) | 28.9 (7.9) | 27.0 (8.2) | 28.4 (8.9)
  Day 21 (n=21, 25, 25, 23) | 29.5 (5.6) | 25.5 (9.3) | 29.7 (7.6) | 27.3 (10.4)

20. Secondary Outcome: Computerized Cognition Assessment: Verbal Memory
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of verbal memory (score range: -60 to 60), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for verbal memory.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 49.4 (4.8) | 48.7 (5.7) | 50.8 (5.9) | 51.5 (4.9)
  Day 21 (n=21, 25, 25, 23) | 52.4 (5.0) | 51.3 (5.2) | 51.2 (6.1) | 50.2 (6.3)

21. Secondary Outcome: Computerized Cognition Assessment: Visual Memory
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of visual memory (score range: -60 to 60), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for visual memory.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 43.0 (6.4) | 43.8 (6.3) | 46.2 (5.8) | 45.3 (6.0)
  Day 21 (n=21, 25, 25, 23) | 46.3 (6.8) | 41.8 (6.7) | 44.8 (7.6) | 45.9 (7.1)

22. Secondary Outcome: Computerized Cognition Assessment: Working Memory
Description: Cognition was assessed by a computerized cognitive testing battery consisting of neuropsychological tests that measure the cognitive domain of working memory (score range: -48 to 48), with a higher score indicating better cognition.
Time Frame: Baseline, Day 21
Population: The ITT population consisted of all participants who were randomized, who received at least one dose of study drug in at least one period, and who had at least one postbaseline computerized cognition efficacy assessment for working memory.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: MK-8777 FD→PBO OR PBO→MK-8777 FD | MK-8777 100mg: MK-8777 FD→PBO OR PBO→MK-8777 FD | Placebo: MK-8777 RD→PBO OR PBO→MK-8777 RD | MK-8777 100-300mg: MK-8777 RD→PBO OR PBO→MK-8777 RD
Number analyzed (Participants) | 27 | 27 | 26 | 32
score on a scale
  BL (n=27, 27, 26, 32) | 9.8 (6.3) | 10.2 (5.0) | 10.0 (5.1) | 9.6 (4.9)
  Day 21 (n=21, 25, 25, 23) | 10.0 (4.1) | 8.5 (5.2) | 10.3 (5.1) | 8.9 (6.0)

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (Up to 12 weeks).
Description: AEs are reported by study drug taken at time of event and not by randomly assigned sequence.
Groups:
- Placebo: Participants receive placebo BID for up to 5 weeks.
- MK-8777 100mg: Participants receive a fixed dose of MK-8777 100 mg BID for up to 3 weeks.
- MK-8777 100-300mg: Participants receive rising doses of MK-8777 100-300 mg BID for up to 3 weeks.
Arm/Group | Placebo | MK-8777 100mg | MK-8777 100-300mg
Serious Adverse Events (participants affected / at risk) | 1/55 | 0/28 | 0/34
Other Adverse Events (participants affected / at risk) | 23/55 | 14/28 | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | MK-8777 100mg (N=28) | MK-8777 100-300mg (N=34)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | MK-8777 100mg (N=28) | MK-8777 100-300mg (N=34)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (4) | 19 (24)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (5) | 15 (17)
Headache (Nervous system disorders) | 7 (7) | 3 (4) | 11 (13)
Somnolence (Nervous system disorders) | 5 (5) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3) | 1 (1)
Thinking abnormal (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less